CLINICAL TRIAL: NCT03948568
Title: A Pragmatic Randomised, Multicentre Trial Evaluating Optimal Timing of Endocrine Therapy and Radiation Therapy in Early-stage Breast Cancer (REaCT-RETT)
Brief Title: Evaluating Optimal Timing of Endocrine Therapy and Radiation Therapy in Early-stage Breast Cancer (REaCT-RETT)
Acronym: REaCT-RETT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 18-02
Record Dates: First submitted 2019-04-18; First posted 2019-05-14 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Early-stage Breast Cancer
Keywords: Radiation Therapy; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Endocrine Therapy and Radiotherapy (Active Comparator): Concurrent endocrine therapy and radiotherapy. Concurrent endocrine therapy will be defined as, the commencement of endocrine therapy around 2 weeks before (a minimum of 1 week before to a maximum of 4 weeks) commencement of radiotherapy and continued throughout radiotherapy.
  Interventions: Combination Product: Endocrine Therapy and Radiotherapy
- Sequential Endocrine Therapy after Radiotherapy (Active Comparator): Sequential endocrine therapy after radiotherapy. Using the pragmatic definition sequential endocrine therapy should commence around 2 weeks (minimum 1 week, maximum 4 weeks) after the last fraction of radiotherapy.
  Interventions: Combination Product: Endocrine Therapy and Radiotherapy

INTERVENTIONS:
Combination Product: Endocrine Therapy and Radiotherapy — Endocrine therapy and radiotherapy administered either concurrently or sequentially
  Other Names: Radiotherapy; Tamoxifen; Letrozole; Anastrozole; Exemestane

SUMMARY:
REaCT-RETT will demonstrate the non-inferiority of concurrent compared to sequential endocrine therapy in patients receiving post-operative radiotherapy for early stage breast cancer.

DETAILED DESCRIPTION:
Clinical equipoise exists around the optimal time to start adjuvant endocrine therapy in patients who will receive post-operative radiotherapy for breast cancer. Patients receive either concurrent or sequential endocrine and radiation therapy, where concurrent therapy consists of endocrine therapy started before, with or during radiotherapy, while sequential treatment is defined as endocrine therapy starting after the completion of radiotherapy. A recent survey of Canadian oncologists showed that the main reason for prescribing sequential endocrine therapy was a concern that concurrent endocrine therapy and radiotherapy would worsen the toxicity of endocrine treatment. This is despite the absence of any clinical trial evidence to support this. Indeed, a recent systematic review by our group was unable to confirm or refute whether increased toxicities, related to the timing of endocrine therapy and radiotherapy actually exist in clinical practice. The investigators are therefore proposing a pragmatic randomised trial to assess whether or not concurrent endocrine therapy and radiotherapy worsens endocrine treatment-related symptoms in an era of modern endocrine and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed early stage, hormone receptor positive breast cancer
* Planned to receive both endocrine therapy and post-operative radiotherapy
* Able to provide verbal consent

Exclusion Criteria:

* Previous endocrine therapy for invasive breast cancer
* Previous radiotherapy for breast cancer in the same breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Endocrine toxicity | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  To measure endocrine toxicity. The Functional Assessment of Cancer Therapy - Endocrine Sub-scale (FACT-ES) is a questionnaire specific to patients with endocrine symptoms and measures the side effects and putative benefits of hormonal treatments given (endocrine therapy) in breast cancer. The FACT-ES questionnaire is comprised of 5 sections; physical well-being (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), functional well-being (7 questions) and additional concerns (19 questions). A total of 46 questions are asked that all contain an answer on a scale range of 0-4, with 0 representing the answer 'not at all' and 4 representing the answer 'very much'. Of the 46 questions asked 31/46 have 'very much' representing the worst answer and the remaining 15/46 have 'very much' representing the best answer.

SECONDARY OUTCOMES:
Radiotherapy toxicity | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  To evaluate the acute and early-moderate late toxicities of radiotherapy in terms of skin toxicity, pneumonitis, and breast pain. This will be recorded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, with breast cosmesis recorded as per the European Organisation for Research and Treatment of Cancer (EORTC) cosmetic rating system for breast cancer. These standardized criteria have been used in a recent Canadian breast radiation randomized trial, RAPID, and the investigators will use a similar template to record any radiation toxicities at different points of time.
Rates of starting endocrine therapy and compliance | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  Rates of starting endocrine therapy, compliance rates, discontinuation rates, along with the reasons for discontinuation.
Direct Estimation of Health Utility Values | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  To measure the patient quality of life using the validated FACT-B questionnaire. The Functional Assessment of Cancer Therapy for Breast Cancer (FACT-B) is a questionnaire that measures multidimensional quality of life in patients with breast cancer. The FACT-B questionnaire is comprised of 5 sections; physical well-being (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), functional well-being (7 questions) and additional concerns (10 questions). A total of 37 questions are asked that all contain an answer on a scale range of 0-4, with 0 representing the answer 'not at all' and 4 representing the answer 'very much'. Of the 46 questions asked 20/37 have 'very much' representing the worst answer and the remaining 17/37 have 'very much' representing the best answer.
Incremental cost-effectiveness ratios | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  Incremental cost-effectiveness ratios (cost per one quality-adjusted life year (QALY) gained and cost per one endocrine toxicity case averted) will be measured using the EQ-5D-5L questionnaire. The EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire consists of two sections; the descriptive system and the visual analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and has 5 levels associated with it (no problems, slight problems, moderate problems, severe problems and extreme problems). The scale range of 1-5 is used for the 5 dimensions where 1 is the best outcome and 5 is the worst outcome. The Visual Analogue scale records the respondent's self-rated health on a vertical, visual scale with endpoints labelled "the best health you can imagine" at the top and "the worst health you can imagine" at the bottom. This ranges 0-100 with 0 being the worst outcome and 100 being the best outcome.
Exploratory analyses on evaluating radiotherapy toxicity | 12 months (+/- 2 weeks) post final fraction of radiotherapy
  Exploratory analyses will be performed evaluating toxicity in patients receiving different types of radiotherapy (i.e. local versus regional radiotherapy). This will be evaluated using data collected on breast volume, seroma size, dose heterogeneity and the time of stimulation and planning.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Bourque, MD, Principal Investigator — Ottawa Hospital Research Institute; Sharon McGee, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada